CLINICAL TRIAL: NCT05755321
Title: From Skin to Brain: Epigenetic Conversion of Skin Fibroblasts Into Neural Stem Cells to Investigate the Impact of Diabetes on Adult Neurogenesis and Neuronal Function
Brief Title: From Skin Fibroblasts to Neural Stem Cells to Investigate in Vitro the Impact of Diabetes on Adult Neurogenesis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Prot 9693/18 ID:1910
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus Type 2 in Obese; Diabetes Mellitus Type 2 in Nonobese; Obesity; Cognitive Dysfunction; Metabolism Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Cognitive Dysfunction; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BMI<25 and T2DM: 10 Subjects with Body Mass Index (BMI) <25 with Type 2 Diabetes Mellitus (T2DM) of both sex.
  Interventions: Other: Skin biopsy
- BMI<25 without T2DM: 10 Subjects with Body Mass Index (BMI) <25 without Type 2 Diabetes Mellitus (T2DM) of both sex.
  Interventions: Other: Skin biopsy
- BMI>30 and T2DM: 10 Subjects with Body Mass Index (BMI) >30 with Type 2 Diabetes Mellitus (T2DM) of both sex.
  Interventions: Other: Skin biopsy
- BMI>30 without T2DM: 10 Subjects with Body Mass Index (BMI) >30 without Type 2 Diabetes Mellitus (T2DM) of both sex.
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — Skin biopsy performed during surgery.

SUMMARY:
Obesity and glucose intolerance or overt diabetes are increasing at an alarming rate in the population, and are bound to become a public health issue and a major cause of disability, loss of independence and high social costs in the near future. A large body of evidence has in recent years highlighted, among the negative effects of overnutrition and glucose dysmetabolism, also an acceleration of cognitive decline and of brain senescence, through cellular (vascular, neuronal, or both) and molecular mechanisms still incompletely clarified. Understanding how overweight and impaired glucose homeostasis negatively affect brain function represents both a major scientific challenge and an avenue to early detection and possibly prevention of this invalidating complication. The aim of this project is to obtain neuronal progenitor-like cells from skin fibroblasts in order to correlate patient-specific metabolism to adult neural stem cell (NSC) and neuronal function in vitro.

DETAILED DESCRIPTION:
* Analysis of skin fibroblasts from normal, obese, lean/diabetic and obese/diabetic individuals and in vitro epigenetic conversion, as revealed by morphological changes, loss of mesenchymal markers and expression of pluripotency genes.
* To re-differentiate patient-derived pluripotent cells into neural progenitor (NP) and to test their proliferative, self-renewal and multilineage differentiation capacity.
* To evaluate neuronal cells derived from patient and control pluripotent cells for a number functional and biochemical parameters (apoptosis/autophagy, mitochondrial potential, reactive oxygen species etc.) relevant to neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with BMI < 25 (normal weight) and BMI > 30 (obese) with or without T2DM with an indication for surgery

Exclusion Criteria:

* Malignant neoplastic diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sexes with BMI < 25 (normal weight) and BMI > 30 (obese) with or without T2DM
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-14 (Estimated)

PRIMARY OUTCOMES:
Fibroblasts culture characterization | About one month to obtain cell cultures from each biopsy. Approximately one month (not necessarily continuous) for in vitro experiments and analyses. Total: 60 days per sample
  To determine whether cells from dysmetabolic individuals are defective (in term of proliferation, senescence, cell death) when compared with control-derived cells
Efficiency of fibroblast epigenetic conversion (gene expression analysis) | The epigenetic conversion protocol requires 25 days, the analysis of gene expression (qRTPCR) approximately 5 days.
  To determine whether cells from dysmetabolic individuals are different in term of epigenetic conversion efficiency when compared with control-derived cells.
Characterization of neural progenitors cells | At the end of the epigenetic conversion, the cell cultures are "blocked" and analysed with biochemistry and molecular biology techniques whose protocols and data analysis require 30 days not necessarily continuous
  To determine whether neural progenitor cell (NPCs) obtained from dysmetabolic individuals are defective (analysis of degenerative features) when compared with control-derived cells.

CONTACTS AND LOCATIONS:
Overall Officials: geltrude mingrone, Principal Investigator — Policlinico A. Gemelli IRCCS
Locations (1):
- Mingrone Geltrude, Roma, Italy